CLINICAL TRIAL: NCT04701203
Title: PaTHway TRIAL: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Trial, With an Open-Label Extension, Investigating the Safety, Tolerability and Efficacy of TransCon PTH Administered Subcutaneously Daily in Adults With Hypoparathyroidism
Brief Title: A Trial Investigating the Safety, Tolerability and Efficacy of TransCon PTH Administered Daily in Adults With Hypoparathyroidism
Acronym: PaTHway
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Bone Diseases A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP-304; 2020-003380-26 (EudraCT Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases
Keywords: Hypoparathyroidism; Parathyroid Hormone; TransCon PTH; PTH(1-34); Prodrug; Sustained Release; Parathyroid Hormone Replacement Therapy; Palopegteriparatide
MeSH Terms: conditions — Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled, parallel group with participants randomized into two treatment groups (3:1): TransCon PTH at a starting dose of 18 mcg/day and titrated to an optimal dose, and placebo for TransCon PTH
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TransCon PTH (Experimental): TransCon PTH at a starting dose of 18 mcg delivered once daily by subcutaneous injection and titrated to an optimal dose
  Interventions: Combination Product: TransCon PTH
- Placebo (Placebo Comparator): Placebo for TransCon PTH delivered once daily by subcutaneous injection
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: TransCon PTH — TransCon PTH drug product is supplied as a solution with a concentration of 0.3 mg PTH(1-34)/mL in a single-patient-use prefilled pen intended for subcutaneous injection.
  Arms: TransCon PTH
Combination Product: Placebo — Placebo is supplied as a solution containing the formulation buffer for TransCon PTH in a single-patient-use prefilled pen intended for subcutaneous injection.
  Arms: Placebo

SUMMARY:
During the first 26 weeks of the trial, participants were randomly assigned to one of two groups: one group received TransCon PTH and one group received placebo. All participants started with study drug at a dose of 18 mcg/day and were individually and progressively titrated to an optimal dose in dose increments of 3 mcg/day. TransCon PTH or placebo were administered as a subcutaneous injection using a pre-filled injection pen. Neither trial participants nor their doctors knew who had been assigned to each group. After the 26 weeks, participants continued in the trial as part of a long-term extension study. During the extension, all participants received TransCon PTH, with the dose adjusted to their individual needs. This was a global trial that was conducted in the United States, Canada, Germany, Denmark, Norway, Italy, and Hungary.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥18 years of age
2. Subjects with postsurgical chronic HP, or auto-immune, genetic, or idiopathic HP for at least 26 weeks. Diagnosis of HP is established based on historic hypocalcemia in the setting of inappropriately low serum PTH levels
3. Requirement for doses of SoC (e.g., calcitriol, alfacalcidol, calcium supplements) at or above a minimum threshold:

   * For countries other than Japan: requirement for a dose of calcitriol ≥0.5 μg/day, or alfacalcidol ≥1.0 μg/day and (elemental) calcium ≥800 mg/day (e.g., calcium citrate, calcium carbonate etc.) for at least 12 weeks prior to Screening. In addition, the dose of calcitriol, or alfacalcidol, or calcium should be stable for at least 5 weeks prior to Screening
   * For Japan: requirement for a dose of calcitriol ≥1.0 μg/day, or alfacalcidol ≥2.0 μg/day for at least 12 weeks prior to Screening. In addition, the dose of calcitriol or alfacalcidol should be stable for at least 5 weeks prior to Screening. In Japan only (due to local practice and dietary patterns), there is no requirement to exceed a minimum dose of calcium supplements
4. Optimization of supplements prior to randomization to achieve the target serum levels of:

   * 25(OH) vitamin D levels of 20-80 ng/mL (49-200 nmol/L) and
   * Magnesium level in the normal range, or just below the normal range and
   * Albumin-adjusted or ionized sCa level in the normal range, or just below the normal range
5. The subject demonstrates a 24-hour uCa excretion of ≥125 mg/24h (on a sample collected within 52 weeks prior to Screening or during the Screening Period)
6. BMI 17- 40 kg/m2 at Screening
7. If ≤25 years of age, radiological evidence of epiphyseal closure based on X-ray of nondominant wrist and hand
8. Thyroid-stimulating hormone (TSH) within normal laboratory limits within the 6 weeks prior to Visit 1; if on suppressive therapy for a history of thyroid cancer, TSH level must be ≥0.2 mIU/mL
9. If treated with thyroid hormone replacement therapy, the dose must have been stable for at least 5 weeks prior to Screening
10. eGFR ≥30 mL/min/1.73 m2 during Screening
11. Able to perform daily subcutaneous self-injections of study drug (or have a designee to perform injections) via a pre-filled injection pen
12. Able and willing to provide written and signed informed consent in accordance with GCP

Exclusion Criteria:

1. Impaired responsiveness to PTH (pseudohypoparathyroidism) which is characterized as PTH-resistance, with elevated PTH levels in the setting of hypocalcemia
2. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis or PTH levels other than HP, such as active hyperthyroidism; Paget disease of bone; severe hypomagnesemia; type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus (HbA1C >9%, documented HbA1C result drawn within 12 weeks prior to Screening is acceptable); severe and chronic liver, or renal disease; Cushing syndrome; multiple myeloma; active pancreatitis; malnutrition; rickets; recent prolonged immobility; active malignancy (other than low-risk well differentiated thyroid cancer or basal cell skin cancer); active hyperparathyroidism; parathyroid carcinoma within 5 years prior to Screening; acromegaly; or multiple endocrine neoplasia types 1 and 2
3. High risk thyroid cancer within 2 years, requiring suppression of TSH <0.2 mIU/mL
4. Use of loop diuretics, phosphate binders (other than calcium supplements), digoxin, lithium, methotrexate, biotin >30 μg/day, or systemic corticosteroids (other than as replacement therapy)
5. Use of thiazide diuretic within 4 weeks prior to the 24-hour urine collection scheduled to occur within 1 week prior to Visit 1
6. Use of PTH-like drugs (whether commercially available or through participation in an investigational trial), including PTH(1-84), PTH(1-34), or other N-terminal fragments or analogs of PTH or PTH-related protein, within 4 weeks prior to Screening
7. Use of other drugs known to influence calcium and bone metabolism, such as calcitonin, fluoride tablets (>0.5 mg/day), strontium, or cinacalcet hydrochloride, within 12 weeks prior to Screening
8. Use of osteoporosis therapies known to influence calcium and bone metabolism, i.e., bisphosphonate (oral or intravenous [IV]), denosumab, raloxifene, or romosozumab therapies within 2 years prior to Screening
9. Non-hypocalcemic seizure disorder with a history of a seizure within 26 weeks prior to Screening
10. Increased risk for osteosarcoma, such as those with Paget's disease of bone or unexplained elevations of alkaline phosphatase, hereditary disorders predisposing to osteosarcoma, or with a prior history of substantial external beam or implant radiation therapy involving the skeleton
11. Pregnant or lactating women
12. Male who has a female partner who intends to become pregnant or is of childbearing potential and is unwilling to use adequate contraceptive methods during the trial
13. Diagnosed drug or alcohol dependence within 3 years prior to Screening
14. Disease processes that adversely affect gastrointestinal absorption, including but not limited to short bowel syndrome, significant small bowel resection, gastric bypass, tropical sprue, active celiac disease, active ulcerative colitis, active Crohn's disease, gastroparesis and AIRE gene mutations with malabsorption
15. Chronic or severe cardiac disease within 26 weeks prior to Screening including but not limited to congestive heart failure, myocardial infarction, severe or uncontrolled arrhythmias, bradycardia (resting heart rate <48 beats/minute, unless chronic and asymptomatic), symptomatic hypotension or systolic BP <80 mm Hg or diastolic <40 mm Hg or poorly controlled hypertension (systolic BP >165 mm Hg or diastolic >95 mm Hg). In the absence of a prior history of hypertension, an isolated BP >165/95 in the setting of white coat hypertension/anxiety may not be exclusionary and a measurement can be repeated prior to randomization
16. Cerebrovascular accident within 5 years prior to Screening
17. Within 26 weeks prior to Screening: acute colic due to nephrolithiasis, or acute gout. Subjects with asymptomatic renal stones are permitted
18. Participation in any other interventional trial in which receipt of investigational drug or device occurred within 8 weeks (or within 5.5 times the half-life of the investigational drug (whichever comes first) prior to Screening
19. Any disease or condition that, in the opinion of the investigator, may require treatment or make the subject unlikely to fully complete the trial, or any condition that presents undue risk from the investigational product or procedures, including treated malignancies that are likely to recur within the approximate 3.5-year duration of the trial
20. Known allergy or sensitivity to PTH or any of the excipients [metacresol, mannitol, succinic acid, NaOH/(HCl)]
21. Likely to be non-compliant with respect to trial conduct
22. Any other reason that in the opinion of the investigator would prevent the subject from completing participation or following the trial schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee D Shu, MD, Study Director — Ascendis Pharma A/S Medical Monitor/Medical Expert
Locations (21):
- United States (9):
  - Ascendis Pharma Investigational Site, San Francisco, California
  - Ascendis Pharma Investigational Site, Chicago, Illinois
  - Ascendis Pharma Investigational Site, Rochester, Minnesota
  - Ascendis Pharma Investigational Site, Reno, Nevada
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Greenville, North Carolina
  - Ascendis Pharma Investigational Site, Austin, Texas
  - Ascendis Pharma Investigational Site, Fort Worth, Texas
  - Ascendis Pharma Investigational Site, Spokane, Washington
- Canada (3):
  - Ascendis Pharma Investigational Site, Halifax, Nova Scotia
  - Ascendis Pharma Investigational Site, Oakville, Ontario
  - Ascendis Pharma Investigational Site, Québec, Quebec
- Denmark (2):
  - Ascendis Pharma Investigational Site, Copenhagen, Capital Region
  - Ascendis Pharma Investigational Site, Aarhus, Central Jutland
- Ascendis Pharma Investigational Site, Dresden, Saxony, Germany
- Hungary (2):
  - Ascendis Pharma Investigational Site, Szeged, Csongrád megye
  - Ascendis Pharma Investigational Site, Budapest
- Italy (3):
  - Ascendis Pharma Investigational Site, Bologna, Emilia-Romagna
  - Ascendis Pharma Investigational Site, Rome, Lazio
  - Ascendis Pharma Investigational Site, Pisa, Piacenza
- Ascendis Pharma Investigational Site, Oslo, Norway

REFERENCES:
- [Derived] Brod M, Pfeiffer KM, Beck JF, Smith A. Measuring treatment impacts on symptoms in adults with hypoparathyroidism: findings from the PaTHway trial. J Patient Rep Outcomes. 2024 Aug 13;8(1):94. doi: 10.1186/s41687-024-00757-1. PMID 39136801
- [Derived] Rejnmark L, Gosmanova EO, Khan AA, Makita N, Imanishi Y, Takeuchi Y, Sprague S, Shoback DM, Kohlmeier L, Rubin MR, Palermo A, Schwarz P, Gagnon C, Tsourdi E, Zhao C, Makara MA, Ominsky MS, Lai B, Ukena J, Sibley CT, Shu AD. Palopegteriparatide Treatment Improves Renal Function in Adults with Chronic Hypoparathyroidism: 1-Year Results from the Phase 3 PaTHway Trial. Adv Ther. 2024 Jun;41(6):2500-2518. doi: 10.1007/s12325-024-02843-8. Epub 2024 Apr 30. PMID 38691316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 84 subjects were randomized and 82 subjects were dosed. Enrollment of subjects occurred in seven countries: Canada, Denmark, Germany, Italy, Hungary, Norway, and the United States.
Pre-assignment Details: A total of 106 subjects were screened and 84 of these met eligibility criteria and were enrolled into the study. Two subjects randomized to TransCon PTH were not treated (1 subject was diagnosed with a recurrence of cancer, and 1 subject withdrew consent). A total of 82 subjects were therefore included in the Intent-to-Treat (ITT) and the Safety analysis populations.
Groups:
- Double Blind: TransCon PTH: TransCon PTH at a starting dose of 18 mcg delivered once daily by subcutaneous injection and titrated to an optimal dose
  TransCon PTH: TransCon PTH drug product is supplied as a solution with a concentration of 0.3 mg PTH(1-34)/mL in a single-patient-use prefilled pen intended for subcutaneous injection.
- Double Blind: Placebo: Placebo for TransCon PTH delivered once daily by subcutaneous injection
  Placebo: Placebo is supplied as a solution containing the formulation buffer for TransCon PTH in a single-patient-use prefilled pen intended for subcutaneous injection.
- Open-Label Extension Period: TransCon PTH: Participants who completed the 26-week double-blind treatment period, continued into the open-label extension period and received treatment with TransCon PTH up to Week 182. All participants received individualized doses of TransCon PTH (allowable dose range: 6 to 60 mcg/day).
Period: Blinded Period (Weeks 0 to 26)
Arm/Group | Double Blind: TransCon PTH | Double Blind: Placebo | Open-Label Extension Period: TransCon PTH
Started | 61 | 21 | 0
Completed | 60 | 19 | 0
Not Completed | 1 | 2 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0
Period: Open-Label Period (Weeks 26 to 182)
Arm/Group | Double Blind: TransCon PTH | Double Blind: Placebo | Open-Label Extension Period: TransCon PTH
Started | 0 | 0 | 79 (Participants who completed the 26-Week double-blind period and entered OLE Period.)
Completed | 0 | 0 | 73
Not Completed | 0 | 0 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 5
Not completed — Pregnancy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TransCon PTH | Placebo | Total
Number analyzed (Participants) | 61 | 21 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.13) | 47.3 (11.43) | 48.6 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 18 | 64
  Male | 15 | 3 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
  White | 57 | 19 | 76
  Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 57 | 18 | 75
  Not Reported | 3 | 1 | 4
  Unknown | 1 | 2 | 3
Height [Mean (Standard Deviation); unit: cm] | 168.22 (8.353) | 166.67 (8.831) | 167.82 (8.450)
Weight [Mean (Standard Deviation); unit: kg] | 77.18 (17.335) | 81.61 (15.631) | 78.31 (16.932)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.27 (5.813) | 29.47 (5.691) | 27.83 (5.828)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Primary Endpoint During the Blinded Period
Description: The primary endpoint was a multi-component endpoint that included the percentage of participants who met the following criteria at 26 weeks of blinded treatment: 1) albumin-adjusted serum calcium measured within 4 weeks prior to and on Week 26 visit within the normal range (8.3 to 10.6 mg/dL), and 2) independence from active vitamin D within 4 weeks prior to Week 26 visit (i.e., all daily standing dose of active vitamin D equal to zero AND use of PRN ≤7 days during the 4 weeks), and 3) independence from therapeutic doses of calcium within 4 weeks prior to Week 26 visit (i.e., average daily standing dose of elemental calcium ≤600 mg AND use of PRN doses on ≤7 days during the 4 weeks), and 4) no increase in prescribed study drug within 4 weeks prior to Week 26 visit.
Time Frame: 26 weeks
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 61 | 21
Percentage of participants | 78.7 [66.3 to 88.1] | 4.8 [0.1 to 23.8]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; For the primary efficacy endpoint, the Cochran-Mantel Haenszel test stratified by etiology of hypoparathyroidism (postsurgical or other) was used to compare the proportion of participants meeting the multi-component primary endpoint in the TransCon PTH versus placebo groups. Participants without week 26 albumin-adjusted serum calcium or with >25% (ie, >7 days) missing diary data of active vitamin D or elemental calcium during the 4 weeks before week 26 were considered non-responders; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Change From Baseline to Week 26 in HPES Symptom - Physical Domain Score
Description: Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Symptom - Physical Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment. The measure uses a scale of 0-100 and values represent the change in scores from baseline. A decrease in HPES score denotes an improvement in hypoparathyroidism disease related physical symptoms.
Time Frame: 26 weeks
Population: The overall number of participants analyzed represents the number of subjects with both baseline and Week 26 visit values available.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 59 | 19
units on a scale | -21.01 [-25.41 to -16.60] | -4.81 [-15.22 to 5.59]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; ANCOVA model with unequal variance was used to analyze the key secondary Endpoints. The change from baseline is variable of interest at week 26 and was included in the model as response variables. Treatment assignment and etiology of hypoparathyroidism were entered as fixed effects and baseline value of the variable of interest was entered as a covariate; Test type: Superiority; p = 0.0038, t-test, 2 sided

3. Secondary Outcome: Change From Baseline to Week 26 in HPES Symptom - Cognitive Domain Score
Description: Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Symptom - Cognitive Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment. The measure uses a scale of 0-100 and values represent the change in scores from baseline. A decrease in HPES score denotes an improvement in hypoparathyroidism disease related cognitive symptoms.
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 59 | 19
units on a scale | -20.49 [-25.67 to -15.31] | -6.16 [-15.92 to 3.60]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0055, t-test, 2 sided

4. Secondary Outcome: Change From Baseline to Week 26 in HPES Impact - Physical Functioning Domain Score
Description: Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Impact - Physical Functioning Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment. The measure uses a scale of 0-100 and values represent the change in scores from baseline. A decrease in HPES score denotes an improvement in physical functioning health-related quality of life.
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 59 | 19
units on a scale | -18.29 [-23.59 to -12.99] | -1.01 [-12.40 to 10.38]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0046, t-test, 2 sided

5. Secondary Outcome: Change From Baseline to Week 26 in HPES Impact - Daily Life Domain Score
Description: Change from baseline in Hypoparathyroidism Patient Experience Scale (HPES) Impact - Daily Life Domain score, a disease-specific patient reported outcome, at 26 weeks of treatment. The measure uses a scale of 0-100 and values represent the change in scores from baseline. A decrease in HPES score denotes an improvement in daily health-related quality of life.
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 59 | 19
units on a scale | -17.65 [-22.39 to -12.91] | -0.36 [-12.19 to 11.46]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0061, t-test, 2 sided

6. Secondary Outcome: Change From Baseline to Week 26 in SF-36 Physical Functioning Subscale Score
Description: Change from baseline in the 36-item Short Form Survey (SF-36) Physical Functioning subscale score, a generic health survey, at 26 weeks of treatment. The Physical Functioning subscale uses a range of 19-57.6 and values represent the change in scores from baseline. An increase in SF-36 score denotes an improvement in physical functioning health-related quality of life.
Time Frame: 26 weeks
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TransCon PTH | Placebo
Number analyzed (Participants) | 59 | 19
units on a scale | 5.29 [3.47 to 7.10] | 0.12 [-4.64 to 4.89]
Statistical Analysis 1: Comparison: TransCon PTH vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0347, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From Week 0 to Week 26 for double-blind treatment period and up to Week 182 for open label extension (OLE)
Description: Analyzed on safety analysis set that included all randomized participants who received at least one dose of trial drug and were analyzed according to actual study treatment received.
Groups:
- Double Blind: TransCon PTH: TransCon PTH at a starting dose of 18 mcg delivered once daily by subcutaneous injection and titrated to an optimal dose during the blinded period
  TransCon PTH: TransCon PTH drug product is supplied as a solution with a concentration of 0.3 mg PTH(1-34)/mL in a single-patient-use prefilled pen intended for subcutaneous injection.
- Double Blind: Placebo: Placebo for TransCon PTH delivered once daily by subcutaneous injection during the blinded period
  Placebo: Placebo is supplied as a solution containing the formulation buffer for TransCon PTH in a single-patient-use prefilled pen intended for subcutaneous injection.
- Total TransCon PTH Period: Participants who completed the 26-week double blind treatment period in placebo and TransCon PTH groups, continued into the open-label extension period and received treatment with TransCon PTH up to Week 182. This period refers to total period of exposure to TransCon PTH. For participants randomized to TransCon PTH at enrollment, the "TransCon PTH Period" was the time from first dose of blinded TransCon PTH until final analysis in OLE period. The TransCon PTH Period for participants randomized to placebo at enrollment was the time from first exposure to TransCon PTH at the time of cross-over from placebo, until final analysis in the OLE period.
Arm/Group | Double Blind: TransCon PTH | Double Blind: Placebo | Total TransCon PTH Period
All-Cause Mortality (participants affected / at risk) | 1/61 | 0/21 | 1/80
Serious Adverse Events (participants affected / at risk) | 5/61 | 2/21 | 20/80
Other Adverse Events (participants affected / at risk) | 50/61 | 20/21 | 72/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: TransCon PTH (N=61) | Double Blind: Placebo (N=21) | Total TransCon PTH Period (N=80)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Endometrial disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind: TransCon PTH (N=61) | Double Blind: Placebo (N=21) | Total TransCon PTH Period (N=80)
Blood thyroid stimulating hormone decreased (Investigations) | 3 | 3 | 11
Hypertension (Vascular disorders) | 3 | 3 | 12
Headache (Nervous system disorders) | 13 | 2 | 19
Paraesthesia (Nervous system disorders) | 12 | 3 | 21
Dizziness (Nervous system disorders) | 4 | 0 | 7
Injection site reaction (General disorders) | 19 | 0 | 20
Fatigue (General disorders) | 9 | 5 | 18
Nausea (Gastrointestinal disorders) | 7 | 2 | 12
Diarrhoea (Gastrointestinal disorders) | 6 | 1 | 7
Constipation (Gastrointestinal disorders) | 4 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 5
Insomnia (Psychiatric disorders) | 4 | 1 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 3 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 2 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 9 | 15
Hypercalcaemia (Metabolism and nutrition disorders) | 5 | 0 | 9
COVID-19 (Infections and infestations) | 1 | 0 | 40
Influenza (Infections and infestations) | 3 | 0 | 8
Nasopharyngitis (Infections and infestations) | 3 | 1 | 7
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 4
Sinusitis (Infections and infestations) | 2 | 0 | 4
Asthenia (General disorders) | 3 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 8
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 7
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 7
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 5
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 8
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 5
Medication error (Injury, poisoning and procedural complications) | 2 | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 4
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 2 | 0 | 7
Palpitations (Cardiac disorders) | 3 | 0 | 9
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 10
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 5
Pneumonia (Infections and infestations) | 0 | 0 | 5
Ear infection (Infections and infestations) | 0 | 0 | 4
Brain fog (Nervous system disorders) | 1 | 1 | 6
Dizziness postural (Nervous system disorders) | 3 | 0 | 4
Non-cardiac chest pain (General disorders) | 1 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 5
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04701203/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT04701203/SAP_001.pdf